CLINICAL TRIAL: NCT01694290
Title: Randomized Controlled Trial Assessing Effectiveness of Chemical Cold Packs Used on Various Skin Surfaces for Cooling Hyperthermic Patients
Brief Title: Chemical Ice Packs for Cooling Hyperthermic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Grant S Lipman, Clinical Associate Professor of Emergency Medicine, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24308
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Heat Stroke, Heat Exhaustion
MeSH Terms: conditions — Heat Stroke; Heat Exhaustion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Chemical Ice packs to neck, groin, axillae (Experimental): Chemical ice packs will be changed out every 9 minutes
  Interventions: Other: Chemical Cold Pack
- Chemical Ice Packs to cheeks, palms, soles (Experimental): Chemical Ice packs will be changed out every 9 minutes
  Interventions: Other: Chemical Cold Pack
- no chemical ice packs (No Intervention)

INTERVENTIONS:
Other: Chemical Cold Pack
  Arms: Chemical Ice Packs to cheeks, palms, soles; Chemical Ice packs to neck, groin, axillae

SUMMARY:
A common tool to cool people in the pre-hospital setting is the chemical ice pack. These are used by athletic trainers, EMS personnel, ER staff, and people in the prehosoital setting.

The ability of these to cool a person has never been quantified, the efficiency and extent of cooling, as well as location of placement of ice packs is purely anecdotal. The purpose of this study is to determine whether strategically placed chemical ice packs will provide benefit to individuals subjected to heat stress.

ELIGIBILITY:
Inclusion Criteria:

* young healthy males > 18 years old with no active medical problems and able to run 10 km.

Exclusion Criteria:

* Active medical problems or inability to exercise for 45 minutes in a heated room.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Core body temperature cooling | 35 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

REFERENCES:
- [Result] Lissoway JB, Lipman GS, Grahn DA, Cao VH, Shaheen M, Phan S, Weiss EA, Heller HC. Novel application of chemical cold packs for treatment of exercise-induced hyperthermia: a randomized controlled trial. Wilderness Environ Med. 2015 Jun;26(2):173-9. doi: 10.1016/j.wem.2014.11.006. Epub 2015 Mar 12. PMID 25771030